CLINICAL TRIAL: NCT01443442
Title: A Single-Center, Masked, Randomized Study Comparing Bepreve (Bepotastine Besilate) 1.5% - H1 Specific Antihistamine vs. Alrex (Loteprednol Etabonate) 0.2% - Corticosteroid in Subjects With Moderate to Severe Allergic Conjunctivitis
Brief Title: Bepreve vs. Alrex in Subjects With Moderate to Severe Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAC-06-11
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Allergic Conjunctivitis
Keywords: Conjunctivitis; Allergic; Bepotastine besilate; Loteprednol etabonate
MeSH Terms: conditions — Conjunctivitis, Allergic; Conjunctivitis | interventions — bepotastine besilate; Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bepreve (Active Comparator): 1.5% bepotastine besilate, drops, twice per day, for two weeks
  Interventions: Drug: bepotastine besilate, 1.5%
- Alrex (Active Comparator): treatment with 0.2 % loteprednol etabonate, drops, four times per day
  Interventions: Drug: Loteprednol etabonate

INTERVENTIONS:
Drug: bepotastine besilate, 1.5% — Topical ocular aqueous formulation, oen drop per instillation, twice per day for 14 days
  Other Names: Bepreve
  Arms: Bepreve
Drug: Loteprednol etabonate — Topical ocular aqueous formulation, one drop per instillation, four times per day for 14 days
  Other Names: Alrex
  Arms: Alrex

SUMMARY:
Allergic conjunctivitis (AC) afflicts approximately 20% of the US population. Typically, patients manifest symptoms in the spring, summer and fall, when airborne allergens are at their peak. Patients may also be afflicted year-round, if sensitive to allergens such as dust mites or pet dander. Signs and symptoms of allergic conjunctivitis are conjunctival hyperemia, ocular itching, conjunctival and eyelid edema, papillary hypertrophy, tearing and burning.

This is a randomized clinical study to evaluate the efficacy of Bepreve® (bepotastine besilate 1.5% ophthalmic solution) compared to Alrex® (loteprednol etabonate 0.2%) in the treatment of moderate to severe allergic conjunctivitis in patient over the age of 18 years. The study will be a two-week study with four visits. Ocular signs (eye redness( and symptoms (itching) will be monitored as outcome variables.

DETAILED DESCRIPTION:
Investigator and Study Center:

Judy Tong, OD Eye Care Center Southern California College of Optometry

Test Product, Dose and Mode of Administration:

Bepreve (bepotastine besilate ophthalmic solution) 1.5% bid ou vs. Alrex (loteprednol etabonate ophthalmic suspension) 0.2% qid ou

Study Title:

A Single-Center, Masked, Randomized Study Comparing Bepreve (bepotastine besilate) 1.5% - H1 Specific Antihistamine vs. Alrex (loteprednol etabonate) 0.2% - Corticosteroid in Subjects with Moderate to Severe Allergic Conjunctivitis

Primary Objective(s):

The primary objective of this study is to compare the efficacy of Bepreve (bepotastine besilate) 1.5% ophthalmic solution compared to Alrex (loteprednol etabonate) 0.2% in the treatment of moderate to severe allergic conjunctivitis in patients over the age of 18 years of age

Study Design:

Interventional, Randomized, Parallel Arm, Investigator Masked

Study Population:

Subjects over the age of 18 years of age with moderate to severe allergic conjunctivitis.

Duration of Treatment: 14 days

Efficacy Assessments: Itching, Bulbar conjunctival injection, Bulbar conjunctival chemosis

Safety Assessments: N/A

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe allergic subjects (≥ 2.5 on a 0.0 to 4.0 itching scale AND

  > grade 2.0 bulbar redness using validated (Efron) scale)
* Must be able to understand and sign an informed consent form that has been approved by the Institutional Review Board (IRB).
* Can comply with instillation of study drug
* Must be able to comply with the visit schedule and other requirements of the study.

Exclusion Criteria:

* Subjects who use daily wear (5-7 days / week, 6-16 hours/day)25 disposable soft hydrogel or silicone hydrogel contact lenses will be included in the study if they have been consistently wearing the same brand and have been using the same care solution for one month or longer. They will be asked to not wear their soft contact lenses to the eligibility visit (three days of no lens wear) and be willing to discontinue lens wear during the two weeks of the study because of the incompatibility of medicated eye drop instillation with contact lens wear and the potential confounding effect of contact lenses and care solutions.
* Active inflammation of the cornea, iris, anterior chamber
* Active or suspected herpetic eye disease (simplex, vaccinia, varicella)
* Active or suspected mycobacterial or acanthamoeba infection
* Active for suspected fungal disorders of the eye
* Persistent and significant dry eye syndrome
* Known allergy, contraindications or hypersensitivity to loteprednol, bepotastine, or its components
* Pregnancy or breast-feeding
* Use of topical eye drops, topical or systemic antihistamines, topical, nasal or systemic corticosteroids, immunosuppressive or immunomodulating agents, decongestants, aspirin, or non-steroidal antiinflammatory (NSAIDs) during the two weeks prior to the study.
* Participation in any other study within 30 days of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Tong, OD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (2):
- United States (2):
  - Eye Car Center, Southern California college of Optometry, Fullerton, California
  - Eye Care Center, Southern Caalifornia College of Optometry, Fullerton, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bepreve | Alrex
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bepreve | Alrex | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Customized [Mean (Standard Deviation); unit: years] | 49.3 (16.3) | 53.0 (13.0) | 51.1 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Itching at 14 Days
Description: Ocular Itching Scale. Scale is 0 - 4 in 0.5 scale unit increments. 0 equals no Itch. 4 equals most severe itch. No calculation details are necessary as the change is calculated as the latest time point minus the earliest time point.
Time Frame: Change from Baseline in Ocular Itching at 14 Days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bepreve | Alrex
Number analyzed (Participants) | 12 | 11
units on a scale | 2.17 (0.53) | 1.82 (0.47)

ADVERSE EVENTS:
Arm/Group | Bepreve | Alrex
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less